CLINICAL TRIAL: NCT01043172
Title: A Phase II Study of Gemcitabine as an Adjuvant Treatment for Cholangiocarcinoma After Surgical Resection
Brief Title: A Study of Gemcitabine as an Adjuvant Treatment for Cholangiocarcinoma After Surgical Resection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Dong-A Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Sang Myung Woo, MD, National Cancer Center, Korea
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GATCO-1
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2018-01

CONDITIONS: Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gemcitabine (Experimental): Gemcitabine : 1000 mg/m2/day D1,8,15 Repeated every 4 weeks 6 cycles
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine : 1000 mg/m2/day D1,8,15 Repeated every 4 weeks 6 cycles
  Other Names: Gemcit

SUMMARY:
The investigators propose to evaluate efficacy and safety of gemcitabine in the adjuvant treatment of cholangiocarcinoma after potentially curative treatment with surgical resection.

DETAILED DESCRIPTION:
Cholangiocarcinoma is a highly fatal disease with poor prognosis. While Cholangiocarcinoma is generally rare in Western countries, it is more common in Korea, with an estimate of 3500 cases diagnosed annually. Currently, surgical resection remains the only potentially curative treatment, but many patients develop recurrence. Thus, effective postoperative adjuvant therapy is required to prolong survival in patients with cholangiocarcinoma. However, no standard postoperative treatment has been established yet.

Among several different new anticancer drugs currently being investigated in the treatment of advanced biliary tract cancer, gemcitabine has generated particular interest. The nucleoside analogue gemcitabine has been reported to be active against advanced unresectable cholangiocarcinoma including cancer of the gallbladder, intrahepatic, and extrahepatic bile duct. So this is expected to be investigated in the adjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects undergoing curative surgical resection for cholangiocarcinoma (including cancer of the gallbladder [except stage I], intrahepatic, and extrahepatic bile duct)
* Histological confirmation is mandatory.
* Age over 18 years old
* Performance status (ECOG scale): 0-2
* Adequate organ functions Hb ≥ 9.0 g/dl ANC: ≥ 1,500/mm3 PLT ≥ 100,000 /mm3 Liver function: Total Bilirubin ≤ 2.0 mg/dl AST / ALT / ALP ≤ 3× upper limit of normal Creatinine ≤ 1.5 ULN
* Patients should sign a written informed consent before study entry.

Exclusion Criteria:

* Tumor type other than adenocarcinoma
* Stage I gallbladder cancer
* Noncurative surgical resection including R2 resection
* Other primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin or prior malignancy treated more than 5 years ago without recurrence)
* Prior systemic therapy (for instance, cytotoxic chemotherapy or active/passive immunotherapy)
* Prior radiotherapy
* Major surgery within 4 weeks prior to study treatment except for surgical resection of cholangiocarcinoma
* Serious illness or medical conditions, as follows; congestive heart failure (NYHA class III or IV) unstable angina or myocardial infarction within the past 6 months, significant arrhythmias requiring medication and conduction abnormality such as over 2nd degree AV block uncontrolled hypertension hepatic cirrhosis(≥ Child class B) interstitial pneumonia, pulmonary adenomatosis psychiatric disorder that may interfere with and/or protocol compliance unstable diabetes mellitus uncontrolled ascites or pleural effusion active infection
* Received any investigational drug or agent/procedure, i.e. participation in another trial within 4 weeks before beginning treatment with study drug
* Pregnant or lactating woman
* Women of child bearing potential not using a contraceptive method
* Sexually active fertile men not using effective birth control during medication of study drug and up to 6 months after completion of study drug if their partners are women of child-bearing potential
* Any patients judged by the investigator to be unfit to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2009-07-20 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Primary objective: To investigate the proportion of patients who are recurrence-free for 2 years | Jan 2010 - Jan 2014 (24 month enrollment, 24 month follow-up)

SECONDARY OUTCOMES:
Time to Recurrence (TTR) Recurrence Free Survival (RFS) QOL | Jan 2010 - Jan 2014 (24 month enrollment, 24 month follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Woo Jin Lee, MD, Principal Investigator — National Cancer Center, Korea
Locations (1):
- National Cancer Center, Goyang-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No